CLINICAL TRIAL: NCT05228470
Title: A PHASE 1B/2, OPEN-LABEL STUDY TO EVALUATE THE SAFETY, PHARMACOKINETICS, PHARMACODYNAMICS, AND EFFICACY OF ELRANATAMAB (PF-06863135) IN CHINESE PARTICIPANTS WITH MULTIPLE MYELOMA WHO ARE REFRACTORY TO AT LEAST ONE PROTEASOME INHIBITOR, ONE IMMUNOMODULATORY DRUG AND ONE ANTI-CD38 ANTIBODY (TRIPLE-CLASS REFRACTORY MM)
Brief Title: A Study of Elranatamab (PF-06863135) in Chinese Participants With Refractory Multiple Myeloma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1071008; NCT05228470 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-01-05; First posted 2022-02-08 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Elranatamab; Myeloma; Multiple Myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma; PF-06863135; BCMA; Bispecific; Bispecific Antibody; BCMA-CD3 Bispecific; MagnetisMM-8
Keywords: Multiple Myeloma; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Hemostatic Disorders; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma; Neoplasms by Histologic Type; Neoplasms; Hemostatic Disorders; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Elranatamab (Experimental): BCMA-CD3 bispecific antibody
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — BCMA-CD3 bispecific antibody
  Other Names: PF-06863135

SUMMARY:
The purpose of this study is to understand the study medicine (called Elranatamab, or PF-06863135) as potential treatment for refractory multiple myeloma. Multiple myeloma is a form of cancer in the bone that forces healthy blood cells to go out. Sometimes, multiple myeloma does not respond to current therapy or quickly progresses, and this is called refractory multiple myeloma.

Elranatamab is a study medicine that target multiple myeloma and activates the human body to fight against this disease. We are seeking Chinese participants to take part in this study. The study will be 2 parts, called part 1b and part 2. In part 1b, participants will receive Elranatamab at 2 steps priming and full dose as a sc (subcutaneous injection) therapy. We will monitor participants' safety and reactions to the study medicine. This will help us understand the dosage of Elranatamab to be used safely.

In part 2 of the study, participants will receive Elranatamab and their multiple myeloma growth will be monitored. This will help us understand if Elranatamab, when used alone, may be a therapy for refractory multiple myeloma. Participants in this part of the study are expected to take part for about 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma (IMWG criteria, Rajkumar et al, 2014)
* Measurable disease, as defined by at least 1 of the following:
* Serum M-protein ≥0.5 g/dL
* Urinary M-protein excretion ≥200 mg/24 hours
* Serum immunoglobulin FLC ≥10 mg/dL (≥100 mg/L) AND abnormal serum immunoglobulin kappa to lambda FLC ratio
* Refractory to at least one IMiD
* Refractory to at least one PI
* Refractory to at least one anti-CD38 antibody
* Relapsed/refractory to last anti-myeloma regimen
* ECOG performance status ≤2
* Adequate BM function characterized by the following:

  1. Absolute neutrophil count ≥1.0 × 10^9/L
  2. Platelets ≥ 25 × 10^9/L
  3. Hemoglobin ≥8 g/dL
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1
* Not pregnant and willing to use contraception

Exclusion Criteria:

* Smoldering multiple myeloma
* Active Plasma cell leukemia
* Amyloidosis
* POEMS syndrome
* Stem cell transplant or active GVHD within 12 weeks prior to enrollment.
* Previous treatment with an anti-BCMA directed therapy
* Impaired cardiovascular function or clinically significant cardiovascular diseases
* Ongoing Grade ≥2 peripheral sensory or motor neuropathy. History of GBS or GBS variants, or history of any Grade ≥3 peripheral motor polyneuropathy.
* Active HBV, HCV, SARS-CoV2, HIV, or any active, uncontrolled bacterial, fungal, or viral infection
* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
* Previous administration with an investigational drug within 30 days or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2025-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- China (15):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shenzhen Second People's Hosptial, Shenzhen, Guangdong
  - Harbin First Hospital, Harbin, Heilongjiang
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Nanjing Drum Tower Hospital,The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shandong Provincial Hospital, Jinan, Shandong
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Beijing Gaobo Boren Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chinese participants with relapsed/refractory multiple myeloma (RRMM), who were refractory to at least 1 proteasome inhibitor (PI), 1 immunomodulatory drug (IMiD), and 1 anti-cluster of differentiation38 monoclonal antibody (anti-CD38 mAB) were included.
Pre-assignment Details: A total of 38 participants were enrolled and assigned to study treatment. Data for only those primary and secondary outcome measures whose analysis is complete and final have been reported. Data for remaining secondary outcome measures will be posted upon completion of analysis at study completion date.
Groups:
- Phase 1b: Participants received subcutaneous (SC) elranatamab with a priming regimen of 12 milligrams (mg) on Cycle 1 Day 1 (C1D1) and 32 mg on Cycle 1 Day 4 (C1D4) followed by 76 mg weekly (QW) thereafter starting from Cycle 1 Day 8. Each cycle was 28 days. If a participant had received QW dosing for at least 6 cycles and had achieved a partial response (PR) or better persisting for at least 2 months, the dose interval was changed to once every 2 weeks (Q2W).
- Phase 2: Participants received SC elranatamab with a priming regimen of 12 mg on C1D1 and 32 mg on C1D4 followed by 76 mg QW thereafter starting from Cycle 1 Day 8. Each cycle was 28 days. If a participant had received QW dosing for at least 6 cycles and had achieved a PR or better persisting for at least 2 months, the dose interval was changed to Q2W.
Period: Overall Study
Arm/Group | Phase 1b | Phase 2
Started | 8 | 30
Completed | 0 | 0
Not Completed | 8 | 30
Not completed — Death | 6 | 11
Not completed — Withdrawal by Subject | 1 | 8
Not completed — Ongoing | 1 | 11

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants enrolled to study who took at least 1 dose of study intervention.
Groups:
- Phase 1b; Phase 2: Participants received SC elranatamab with a priming regimen of 12 mg on C1D1 and 32 mg on C1D4 followed by 76 mg QW thereafter starting from Cycle 1 Day 8.
- Total: Total of all reporting groups
Arm/Group | Phase 1b | Phase 2 | Total
Number analyzed (Participants) | 8 | 30 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (12.19) | 62.3 (7.53) | 60.7 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 16
  Male | 4 | 18 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 30 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 30 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: Grade(G)4 neutropenia >5 day; febrile neutropenia (absolute neutrophil count [ANC] <1000/millimeter cube (mm^3) with single temperature >38.3 degree Celsius (deg C) or sustained temp>=38 deg C for >1 hour(H); G>=3 neutropenia with infection; G4 thrombocytopenia (unless baseline count >=25,000/mm^3 and <50,000/mm^3, in which case G4 thrombocytopenia to be accompanied by >=G2 bleeding); Platelet count <10,000/mm^3; G3 thrombocytopenia with >=G2 bleeding; G>=4 AE; G3 cytokine release syndrome(CRS) except CRS not maximally treated/improved to <=G1 within 48H; G3 AE except AE attributed to CRS, G3 nausea,vomiting,diarrhea improved to G<=2 within 72H after medical management, G3 fatigue <1 week, G3 AE recovered to baseline/G1 within 5 day; confirmed drug-induced liver injury; G3-4 laboratory (lab) abnormality except G3-4 lab abnormality improved to G<=2 within 72H after medical management & without sequelae;G3 injection site reaction; G2/other clinically important AE may be considered DLT.
Time Frame: Cycle 1 (28 days)
Population: DLT evaluable analysis set included all participants enrolled to Phase 1b part and who had a DLT in the DLT observation period or completed the DLT observation period without DLT. Participants without DLTs and without the minimum required exposure for reasons other than treatment-related toxicity were not evaluable for DLTs and were replaced.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Objective Response Rate (ORR) by Blinded Independent Central Review (BICR) as Per International Myeloma Working Group (IMWG) Criteria
Description: ORR: Percentage of participants with best overall response of confirmed stringent complete response (sCR), CR, very good partial response (VGPR) or PR per IMWG criteria. sCR: CR & normal serum free light chain (sFLC) ratio & absence of clonal cells in BMB/BMA by IH, IF, or flow cytometry. CR: negative immunofixation on serum & urine, disappearance of any soft tissue plasmacytoma & <5% plasma cells in BMA, if disease measurable by sFLC only, preceding criteria plus normal sFLC ratio. VGPR: Serum & urine M-protein detectable by immunofixation but not on electrophoresis; or >=90% reduction in serum M-protein & urine M-protein level <100mg/24h. PR: >=50% reduction in serum M-protein & reduction in 24h urinary M-protein by >=90% or <200 mg/24h. If serum & urine M-protein were unmeasurable, VGPR & PR: >=90% & >=50% decrease in difference respectively between involved & uninvolved sFLC levels & if present at baseline, >=90% & >=50% reduction in soft tissue plasmacytomas' size.
Time Frame: From date of first dose until confirmed disease progression, death, start of new anticancer therapy, whichever occurred first (approximately up to 16 months)
Population: The primary analysis of ORR as planned per protocol included participants who started with the recommended phase 2 dose [RP2D] (including the participants from both Phase 1b and Phase 2 parts). Safety analysis set included all enrolled participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase 1b + Phase 2: Participants received SC elranatamab with a priming regimen of 12 mg on C1D1 and 32 mg on C1D4 followed by 76 mg QW thereafter starting from Cycle 1 Day 8.
Arm/Group | Phase 1b | Phase 2 | Phase 1b + Phase 2
Number analyzed (Participants) | 8 | 30 | 38
Percentage of participants | 37.5 [8.5 to 75.5] | 53.3 [34.3 to 71.7] | 50.0 [33.4 to 66.6]
Statistical Analysis 1: Comparison: Phase 1b + Phase 2; Test type: Other — Null hypothesis of ORR by BICR was 30%; p = 0.0076, Exact binomial test

3. Secondary Outcome: Duration of Response (DOR) as Per IMWG Criteria by BICR
Description: DOR: Time from first documentation of objective response subsequently confirmed, until first documentation of confirmed PD or death due to any cause, whichever occurred first. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5g/dL]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200mg/24h]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved sFLC levels [absolute increase >10mg/dL]; in participants without measurable serum, urine M-protein levels & involved sFLC levels: bone marrow plasma-cell % irrespective of baseline status [absolute increase >=10%]; appearance of new lesion,>=50% increase from nadir in SPD of >1 lesion, or >=50% increase in longest diameter of previous lesion >1cm in short axis; >=50% increase in circulating plasma cells [>=200cells/μL] if this is the only measure of disease.
Time Frame: From first documentation of objective response subsequently confirmed until confirmed PD or death due to any cause, or start of new anticancer therapy, whichever occurred first, or censoring (up to approximately 37 months)
Reporting Status: Not Posted, anticipated posting 2026-09

4. Secondary Outcome: Duration of Response (DOR) as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 3
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2026-09

5. Secondary Outcome: Complete Response Rate (CRR) as Per IMWG Criteria by BICR
Description: CRR: Percentage of participants with BOR of confirmed sCR/CR per IMWG criteria. sCR: CR & normal serum free light chain (sFLC) ratio & absence of clonal cells in BMB/BMA by IH, IF, or flow cytometry. CR: negative immunofixation on serum & urine, disappearance of any soft tissue plasmacytoma & <5% plasma cells in BMA, if disease measurable by sFLC only, preceding criteria plus normal sFLC ratio.
Time Frame: From date of first dose until confirmed disease progression, death, start of new anticancer therapy, whichever occurred first (up to approximately 37 months)
Reporting Status: Not Posted, anticipated posting 2026-09

6. Secondary Outcome: Complete Response Rate (CRR) as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 5
Time Frame: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2026-09

7. Secondary Outcome: Objective Response Rate (ORR) as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 2
Time Frame: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2026-09

8. Secondary Outcome: Duration of Complete Response (DOCR) as Per IMWG Criteria by BICR
Description: DOCR: Time from first documentation of sCR/CR subsequently confirmed, until first documentation of confirmed PD or death due to any cause, whichever occurred first. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5g/dL]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200mg/24h]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved sFLC levels [absolute increase >10mg/dL]; in participants without measurable serum, urine M-protein levels & involved sFLC levels: bone marrow plasma-cell % irrespective of baseline status [absolute increase >=10%]; appearance of new lesion,>=50% increase from nadir in SPD of >1 lesion, or >=50% increase in longest diameter of previous lesion >1cm in short axis; >=50% increase in circulating plasma cells [>=200cells/μL] if this is the only measure of disease.
Time Frame: From first documentation of sCR/CR subsequently confirmed until confirmed PD or death due to any cause, or start of new anticancer therapy, whichever occurred first, or censoring (up to approximately 37 months)
Reporting Status: Not Posted, anticipated posting 2026-09

9. Secondary Outcome: Duration of Complete Response (DOCR) as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 8
Time Frame: From the first documentation of sCR/CR, until confirmed PD per IMWG criteria, or death due to any cause, whichever occurred first (up to approximately 37 months)
Reporting Status: Not Posted, anticipated posting 2026-09

10. Secondary Outcome: Progression Free Survival (PFS) as Per IMWG Criteria by BICR
Description: PFS was defined as the time from the date of first dose until confirmed PD or death due to any cause, whichever occurred first. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5g/dL]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200mg/24h]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved sFLC levels [absolute increase >10mg/dL]; in participants without measurable serum, urine M-protein levels & involved sFLC levels: bone marrow plasma-cell % irrespective of baseline status [absolute increase >=10%]; appearance of new lesion,>=50% increase from nadir in SPD of >1 lesion, or >=50% increase in longest diameter of previous lesion >1cm in short axis; >=50% increase in circulating plasma cells [>=200cells/μL] if this is the only measure of disease.
Time Frame: From date of first dose until confirmed PD or death due to any cause, or start of new anticancer therapy, whichever occurred first, or censoring (up to approximately 37 months)
Reporting Status: Not Posted, anticipated posting 2026-09

11. Secondary Outcome: Progression Free Survival (PFS) as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 10
Time Frame: as for outcome 10
Reporting Status: Not Posted, anticipated posting 2026-09

12. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from date of first dose until death due to any cause.
Time Frame: From the date of first dose until death due to any cause. Participants not known to have died were censored on the date of last known alive (up to approximately 37 months)
Reporting Status: Not Posted, anticipated posting 2026-09

13. Secondary Outcome: Time-to-Response (TTR) as Per IMWG Criteria by BICR
Description: TTR was defined, for participants with an objective response per IMWG criteria, as the time from the date of first dose to the first documentation of objective response that was subsequently confirmed.
Time Frame: From date of first dose until confirmed disease progression, death, start of new anticancer therapy, whichever occurs first (approximately up to 16 months)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study intervention. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1b | Phase 2 | Phase 1b + Phase 2
Number analyzed (Participants) | 3 | 16 | 19
Months | 2.04 [1.15 to 4.73] | 1.45 [0.95 to 5.52] | 1.51 [0.95 to 5.52]

14. Secondary Outcome: Time-to-Response (TTR) as Per IMWG Criteria by Investigator Assessment
Description: as for outcome 13
Time Frame: From date of first dose until confirmed disease progression, death, start of new anticancer therapy, whichever occurs first (up to approximately 37 months)
Reporting Status: Not Posted, anticipated posting 2026-09

15. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate Per IMWG Sequencing Criteria
Description: MRD negativity rate was the percentage of participants with CR/sCR and with negative MRD per IMWG sequencing criteria.
Time Frame: as for outcome 5
Reporting Status: Not Posted, anticipated posting 2026-09

16. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE), Serious TEAEs, Treatment Related TEAEs, Serious Treatment Related TEAEs as Graded by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0
Description: AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to study intervention. An SAE was defined as any untoward medical occurrence that, at any dose resulted in any of the following outcomes: death; life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; or that was considered as an important medical event. An AE was considered treatment-emergent if it occurred from the first dose of the study intervention until 90 days after the last dose or the day before starting a new anticancer therapy, whichever occurred first. CTCAE version 5.0 Grade 1: mild; Grade 2: moderate; Grade 3: severe or clinically significant; Grade 4: life-threatening; Grade 5: death.
Time Frame: From the date of first dose up to 90 days after last dose or new anticancer therapy whichever occurred first (up to approximately 37 months)
Reporting Status: Not Posted, anticipated posting 2026-09

17. Secondary Outcome: Number of Participants With Cytokine Release Syndrome (CRS) Graded According to American Society for Transplantation and Cellular Therapy (ASTCT) Criteria
Description: ASTCT CRS Grading: Grade 1: temperature >=38°C without hypotension or hypoxia; Grade 2: temperature >=38°C with hypotension not requiring vasopressors, and/or hypoxia requiring low-flow nasal cannula, facemask or blow-by; Grade 3: temperature >=38°C with hypotension requiring a vasopressor with or without vasopressin and/or hypoxia requiring high-flow nasal cannula, facemask, nonrebreather mask, or Venturi mask; Grade 4: temperature >=38°C with hypotension requiring multiple vasopressors (excluding vasopressin) and/or hypoxia requiring positive pressure (eg, continuous positive airway pressure [CPAP], bilevel positive airway pressure [BiPAP], intubation and mechanical ventilation); Grade 5: death
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-09

18. Secondary Outcome: Number of Participants With Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) Graded According to ASTCT Criteria
Description: ICANS Grade 1: immune effector cell encephalopathy (ICE) score 7-9, participant awakens spontaneously; Grade 2: ICE score 3-6, participant awakens to voice; Grade 3: ICE score 0-2, participant awakens only to tactile stimulus, any clinical seizure focal or generalized that resolved rapidly or nonconvulsive seizures on electroencephalography that resolve with intervention or focal/local edema on neuroimaging; Grade 4: ICE score 0 (participant is unarousable and unable to perform ICE), participant unarousable or requires vigorous or repetitive tactile stimuli to arouse, life-threatening prolonged seizure (>5 min), repetitive clinical or electrical seizures without return to baseline in between, deep focal motor weakness, diffuse cerebral edema on neuroimaging; decerebrate/decorticate posturing; cranial nerve VI palsy; papilledema, Cushing's triad; Grade 5: death. ICE: measures alterations in speech, orientation, handwriting, attention and receptive aphasia.
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2026-09

19. Secondary Outcome: Maximum Serum Concentration (Cmax) of Free Elranatamab
Time Frame: Cycle 1: Pre-dose, 6 hours post-dose on Day 1, 24, 48 hours post-dose, Day 4: pre-dose, 24 hour post-dose, Day 8 pre-dose, 6 hours post-dose, Day 15,22: pre-dose, Cycles 2, 3 ,4,7: pre-dose (1 cycle =28 days)
Population: Pharmacokinetic (PK) parameter analysis set included all participants enrolled and treated who had at least 1 of the PK parameters of primary interest in the single dose and/or multiple-dose PK part. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Phase 1b | Phase 2 | Phase 1b + Phase 2
Number analyzed (Participants) | 7 | 6 | 13
Microgram per milliliter | 0.8762 (66) | 0.8039 (24) | 0.8420 (48)

20. Secondary Outcome: Time To Maximum Serum Concentration (Tmax) of Free Elranatamab
Time Frame: as for outcome 19
Population: PK parameter analysis set included all participants enrolled and treated who had at least 1 of the PK parameters of primary interest in the single dose and/or multiple-dose PK part. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Phase 1b | Phase 2 | Phase 1b + Phase 2
Number analyzed (Participants) | 7 | 6 | 13
Days | 7.00 [3.93 to 9.97] | 8.00 [6.94 to 11.0] | 7.00 [3.93 to 11.0]

21. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Time of Last Measurable Concentration (AUClast) of Free Elranatamab
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*day per milliliter
Arm/Group | Phase 1b | Phase 2 | Phase 1b + Phase 2
Number analyzed (Participants) | 7 | 6 | 13
Microgram*day per milliliter | 3.482 (74) | 3.864 (37) | 3.653 (56)

22. Secondary Outcome: Serum Concentration of Free Elranatamab
Time Frame: Up to 37 months
Reporting Status: Not Posted, anticipated posting 2026-09

23. Secondary Outcome: Percentage of Participants With Positive Anti-Drug Antibody (ADA) and Neutralizing Antibodies (NAb) Against Elranatamab
Time Frame: From the date of first dose up to 37 months
Reporting Status: Not Posted, anticipated posting 2026-09

24. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life of Cancer Participants Core Module (EORTC QLQ-C30)
Description: EORTC QLQ-C30 contains 30 items and is composed of both multi-item scales and single-item measures. These include 5 functional scales (physical, role, emotional, cognitive and social functioning), 3 symptom scales (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/QoL scale. All the scales and single-item measures range in score from 0 to 100. Higher scores on the functional scales represent higher levels of functioning. Higher scores on the global health status/quality of life scale represent higher health status/quality of life. Higher scores on symptom scales/items represent a greater presence of symptoms.
Time Frame: Baseline and up to 37 months
Reporting Status: Not Posted, anticipated posting 2026-09

25. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Myeloma-Specific Module (EORTC QLQ-MY20)
Description: EORTC MY20 is a myeloma-specific module developed by the EORTC group specifically to assess quality of life in participants with multiple myeloma. It contains 20 items which can be grouped into a disease symptom subscale (6 items), side effects of treatment subscale (10 items), body image (1 item) and future perspective subscale (3 items). All transformed scale scores range from 0 to 100 with higher scores indicating worse symptoms (Disease Symptoms and Side Effects of Treatment) or better support/functioning (Future Perspective and Body Image).
Time Frame: Baseline and up to 37 months
Reporting Status: Not Posted, anticipated posting 2026-09

26. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire- Chemotherapy-Induced Peripheral Neuropathy (EORTC QLQ CIPN20)
Description: EORTC QLQ CIPN20 is a module developed by the EORTC group to assess chemotherapy-induced peripheral neuropathy. It contains 20 items which can be grouped into a sensory subscale (9 items), motor subscale (8 items) and autonomic subscale (3 items). Sensory scale scores range from 1 to 36, motor scale scores range from 1 to 32, and autonomic scale scores range from 1 to 12 for men and 1-8 for women (erect dysfunction item excluded). Higher scores indicate worse neuropathy.
Time Frame: Baseline and up to 37 months
Reporting Status: Not Posted, anticipated posting 2026-09

27. Secondary Outcome: Change From Baseline in EuroQol Five Dimensions Questionnaire (EQ-5D) Index Score and in EQ-5D Visual Analogue Score (VAS) (EQ-VAS)
Description: The EQ-5D is a 6-item questionnaire with 2 components, a Health State Profile which has individuals rate their level of problems in 5 areas (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), and a VAS in which patients rate their overall health status from 0 (worst imaginable) to 100 (best imaginable). Overall scores range from 0 to 1, with lower scores representing higher levels of dysfunction. EQ-VAS records the participant's self-rated health on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline and up to 37 months
Reporting Status: Not Posted, anticipated posting 2026-09

ADVERSE EVENTS:
Time Frame: AEs: From the date of first dose up to 90 days after last dose or new anticancer therapy whichever occurred first (approximately up to 16 months)
Description: Same event may appear as both non-SAE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set evaluated. All-Cause Mortality:total number of deaths during study,from first dose of study drug and up to end of study are reported for all treated participants and included deaths which occurred after 90 days post last dose of study drug.
Arm/Group | Phase 1b | Phase 2 | Phase 1b + Phase 2
All-Cause Mortality (participants affected / at risk) | 6/8 | 13/30 | 19/38
Serious Adverse Events (participants affected / at risk) | 6/8 | 23/30 | 29/38
Other Adverse Events (participants affected / at risk) | 8/8 | 30/30 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b (N=8) | Phase 2 (N=30) | Phase 1b + Phase 2 (N=38)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Death (General disorders) | 0 | 2 | 2
Fatigue (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 1 | 2
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 1 | 2 | 3
COVID-19 pneumonia (Infections and infestations) | 0 | 2 | 2
Erysipelas (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Haematological infection (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Herpes zoster meningoencephalitis (Infections and infestations) | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 3 | 12 | 15
Sepsis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Globulins decreased (Investigations) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1
Intracranial mass (Nervous system disorders) | 0 | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b (N=8) | Phase 2 (N=30) | Phase 1b + Phase 2 (N=38)
Anaemia (Blood and lymphatic system disorders) | 6 | 20 | 26
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2 | 2
Hypoglobulinaemia (Blood and lymphatic system disorders) | 1 | 3 | 4
Leukopenia (Blood and lymphatic system disorders) | 7 | 20 | 27
Lymphopenia (Blood and lymphatic system disorders) | 4 | 16 | 20
Neutropenia (Blood and lymphatic system disorders) | 7 | 22 | 29
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 19 | 27
Cardiac failure (Cardiac disorders) | 1 | 2 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 3 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 2 | 2
Conjunctival hyperaemia (Eye disorders) | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 5
Aphthous ulcer (Gastrointestinal disorders) | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 4 | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 8 | 11
Frequent bowel movements (Gastrointestinal disorders) | 0 | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2
Mouth ulceration (Gastrointestinal disorders) | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 3 | 3 | 6
Vomiting (Gastrointestinal disorders) | 3 | 2 | 5
Asthenia (General disorders) | 1 | 10 | 11
Chest discomfort (General disorders) | 1 | 2 | 3
Fatigue (General disorders) | 3 | 1 | 4
Injection site reaction (General disorders) | 1 | 9 | 10
Oedema peripheral (General disorders) | 2 | 1 | 3
Pain (General disorders) | 0 | 3 | 3
Pyrexia (General disorders) | 4 | 9 | 13
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 3 | 4
Hepatic steatosis (Hepatobiliary disorders) | 0 | 2 | 2
Cytokine release syndrome (Immune system disorders) | 3 | 15 | 18
COVID-19 (Infections and infestations) | 2 | 20 | 22
Cytomegalovirus infection (Infections and infestations) | 0 | 3 | 3
Herpes zoster (Infections and infestations) | 0 | 3 | 3
Infection (Infections and infestations) | 0 | 2 | 2
Pneumonia (Infections and infestations) | 5 | 10 | 15
Sinusitis (Infections and infestations) | 1 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 8
Urinary tract infection (Infections and infestations) | 1 | 2 | 3
Alanine aminotransferase increased (Investigations) | 0 | 6 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 7 | 7
Bile acids increased (Investigations) | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 7 | 7
Blood bilirubin increased (Investigations) | 1 | 4 | 5
Blood creatinine increased (Investigations) | 1 | 1 | 2
Blood glucose increased (Investigations) | 0 | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 3 | 8 | 11
Blood urea increased (Investigations) | 2 | 0 | 2
C-reactive protein increased (Investigations) | 1 | 1 | 2
CD19 lymphocytes decreased (Investigations) | 1 | 1 | 2
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 8 | 8
Globulins decreased (Investigations) | 1 | 2 | 3
Interleukin level increased (Investigations) | 3 | 4 | 7
Neutrophil count increased (Investigations) | 1 | 1 | 2
Procalcitonin increased (Investigations) | 0 | 2 | 2
SARS-CoV-2 test positive (Investigations) | 2 | 20 | 22
Serum ferritin increased (Investigations) | 1 | 1 | 2
T-lymphocyte count increased (Investigations) | 1 | 1 | 2
Weight decreased (Investigations) | 1 | 6 | 7
Decreased appetite (Metabolism and nutrition disorders) | 1 | 7 | 8
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 3 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 6 | 8
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 9 | 10
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 8 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 5 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 12 | 14
Hypochloraemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 16 | 21
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 8 | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 3 | 5
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 2 | 3
Headache (Nervous system disorders) | 2 | 1 | 3
Insomnia (Psychiatric disorders) | 2 | 7 | 9
Renal failure (Renal and urinary disorders) | 0 | 2 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hypotension (Vascular disorders) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT05228470/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT05228470/SAP_001.pdf